CLINICAL TRIAL: NCT06474390
Title: Validation of a Medical-grade Wearable Device with Interpretable Artificial Intelligence System for the Obstructive Sleep Apnea-hypopnea Syndrome (OSAHS) Evaluation
Brief Title: TipTraQ Home Sleep Test Validation Study, VGH
Status: Recruiting | Type: Observational
Sponsor: PranaQ Pte. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: TipTraQ validation VGH
Record Dates: First submitted 2024-06-13; First posted 2024-06-25 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; home sleep test; wearble device
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A validation study has been designed to assess the performance of a home sleep test device, TipTraQ, for screening sleep apnea. The study involves participants wearing the TipTraQ device on their fingertip during a traditional sleep test, known as polysomnography (PSG), conducted in a sleep center. The performance of the device will then be evaluated by comparing the results from the TipTraQ system with those from the traditional sleep test.

DETAILED DESCRIPTION:
This clinical study is designed to validate TipTraQ, a new sleep screening device developed by PranaQ, for the detection of Sleep Breathing Disorders (SBD), including obstructive sleep apnea-hypopnea syndrome (OSAHS). Given the high prevalence of undiagnosed OSAHS and the cumbersome nature of traditional polysomnography (PSG) - which involves multiple sensors and specialist interpretation - there is a pressing need for more accessible screening tools. TipTraQ aims to meet this need through a wearable device that utilizes photoplethysmography (PPG) and an accelerometer to monitor essential physiological parameters during sleep. This information is then analyzed by an interpretable artificial intelligence (AI) system to estimate key indicators of sleep health such as SpO2, total sleep time (TST), oxygen desaturation index (ODI), and apnea-hypopnea index (AHI).

The study is open-label and non-randomized, planning to recruit 125 subjects. Participants will use the TipTraQ device alongside a companion mobile app, with data analysis supported by AI technology hosted on a cloud server. The primary goal is to assess the accuracy of the TipTraQ system by comparing its output against the gold standard PSG annotations made by sleep experts.

This initiative represents a significant step towards simplifying and democratizing the screening process for sleep disorders, potentially enabling early detection and treatment for a larger segment of the population, thus mitigating personal health risks and broader societal impacts of undiagnosed SBD.

ELIGIBILITY:
Inclusion Criteria:

Subjects from the age of 20 and older that have an indication for an in-lab PSG study in the Duke University Hospital. The subject should be able to understand the study and sign the informed consent before being enrolled in the study. During the study period, the subject can withdraw from the study anytime.

Exclusion Criteria:

Subjects with the following medical conditions will be excluded from this study:

1. Heart transplant
2. Heart failure, New Youk Heart Association (NYHA) classification III or IV
3. Chronic Obstructive Lung Disease, Global Initiative for Chronic Obstructive Lung Disease (GOLD) categorization 3 or 4
4. Chronic opioid medication user Devastating Severe strokes, with the modified Rankin score (mRS)≥4
5. Tracheostomy
6. Incapable of comprehending and signing the informed consent and questionnaires, including but not limited to subjects with severe Alzheimers, unconscious by head trauma, or of someone with limited mental capacity Cannot correctly follow the order to use the TipTraQ device

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy or people who has indication to conduct polysomnography (PSG).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen Desaturation Index(ODI) | From the start of a single polysomnography study to the end of the recording. Time range from 4hour up to 10 hour.
  Average desaturation episodes with a decrease in the oxygen saturation of ≥4% or 3% per hour
Apnea Hypopnea Index(AHI) | From the start of a single polysomnography study to the end of the recording. Time range from 4hour up to 10 hour.
  The combined average number of apneas and hypopneas that occur per hour of sleep
Total Sleep Time(TST) | From the start of a single polysomnography study to the end of the recording. Time range from 4hour up to 10 hour.
  Total sleep time during the polysomnography (PSG)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The study collects mostly physiological signal data, not suitable for IPD